CLINICAL TRIAL: NCT02560402
Title: Relation Between Renal Resistive Index, Glomerular Hyperfiltration and Hyperdynamic Circulation in Critically Ill Patients With Trauma or Sepsis.
Brief Title: The Relation Between the Renal Resistive Index and Glomerular Hyper Filtration
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M. Oudemans-van Straaten, MD, PhD, Prof. Dr., Amsterdam UMC, location VUmc
Other Study IDs: METC-2014.563
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Trauma; Sepsis
Keywords: Glomerular hyperfiltration; Renal Resistive Index (RRI)
MeSH Terms: conditions — Wounds and Injuries; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with sepsis or trauma: Adult patients, admitted to the intensive or medium care unit with sepsis or trauma

SUMMARY:
Aim of the present study is to determine whether

1. RRI can predict glomerular hyperfiltration;
2. glomerular hyperfiltration is associated with low renal resistive index;
3. glomerular hyperfiltration/low RRI are associated with accelerated flow in the sublingual microcirculation;
4. glomerular hyperfiltration/low RRI are related to fluid status as quantified with bioimpedance analysis.

DETAILED DESCRIPTION:
Apart from acute kiddney injury (AKI), critically ill patients with sepsis or trauma can also exhibit glomerular hyperfiltration (2-4). Glomerular hyperfiltration is not easily recognized, because the decrease in serum creatinine is a late manifestation and generally interpreted as normal renal function. Glomerular hyperfiltration may have clinical consequences, because it leads to augmented renal clearance of water soluble drugs. This is especially relevant for antibiotics, because augmented clearance can lead to underdosing and therapeutic failure (5-9). Patients with glomerular hyperfiltration are generally younger patients with less severe disease (3) and often exhibit a hyperdynamic circulation. The mechanism of glomerular hyperfiltration is poorly understood. High catecholamine release with increased renal blood flow could play a role. Direct measurement of renal blood flow is not available in daily clinical practice.

Nowadays, the investigators can measure Renal Resistive Index (RRI) using renal Doppler ultrasound. The RRI is a sonographic index assessing resistance of the intrarenal arcuate or interlobar arteries and is normally used to assess renal arterial disease. The method has now become available at the bedside in the intensive care unit. RRI is calculated as: (peak systolic velocity - end diastolic velocity)/peak systolic velocity. Normal values are between 0.60 and 0.70. A mean value of 0.72 has been found in critically ill patients admitted to the intensive care unit (personal data).

The investigators hypothesize that high glomerular filtration rate as measured with creatinine clearance is associated with a low renal resistive index and accelerated microvascular blood flow.

To prove or reject this hypothesis, the following study measurements will be performed in critically ill patients with sepsis or trauma:

1. Renal ultrasound to measure renal resistive index (RRI) After visualising the kidney in ultrasound mode, checking for (chronic) renal damage, an arcuate or interlobar artery will be localized and three successive Doppler measurements at different positions in the kidney (high, middle and low) will be performed. This will be repeated 3 times in each kidney. So a total number of 9 RRI values will be obtained in each kidney.
2. Sublingual microcirculation using Sidestream Dark Field imaging (SDF) After removal of secretions with a gauze, the device will be applied below the tongue and three sequences of about 20 seconds from adjacent areas will be recorded and stored. The investigators will measure the perfused vessel density (PVD), the proportion of perfused vessels (PPV) and the microvascular flow index (MFI) for small vessels. Each image will be divided into four quadrants, and the predominant type of flow (0 = absent, 1 = intermittent, 2 = sluggish, 3 = normal, 4 = high) will be evaluated in each quadrant. The mean of the four quadrants will be used for analysis.
3. To assess fluid status, Bioelectrical impedance analysis (BIA) will be performedusing the Akern BIA 101 device.

BIA measures Resistance (R) and Reactance (Xc) reflecting extracellulair (R) and cellular (Xc) resistance to an alternating current of 400 μA with afrequency of 50 kHz. In previous studies the investigators found that (changes in) R are highely correlation with (changes in) fluid status.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the intensive or medium care unit
* Sepsis or trauma
* Age > 18 years

Exclusion Criteria:

Patients

* with chronic renal insufficiency (eGFR < 30 ml)
* with renal transplant kidney
* on chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, admitted to the intensive or medium care unit with sepsis or trauma
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Renal Resistive Index (RRI) | 1 week

SECONDARY OUTCOMES:
4-h Creatinine clearance | 1 week
Microvascular flow index of the sublingual microcirculation | 1 week
Resistance, as measured with bioimpedance as a marker of fluid status. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Heleen M. Oudemans, Prof. Dr., Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellomo R, Kellum JA, Ronco C. Acute kidney injury. Lancet. 2012 Aug 25;380(9843):756-66. doi: 10.1016/S0140-6736(11)61454-2. Epub 2012 May 21. PMID 22617274
- [Background] Udy A, Boots R, Senthuran S, Stuart J, Deans R, Lassig-Smith M, Lipman J. Augmented creatinine clearance in traumatic brain injury. Anesth Analg. 2010 Dec;111(6):1505-10. doi: 10.1213/ANE.0b013e3181f7107d. Epub 2010 Nov 3. PMID 21048095
- [Background] Udy AA, Roberts JA, Shorr AF, Boots RJ, Lipman J. Augmented renal clearance in septic and traumatized patients with normal plasma creatinine concentrations: identifying at-risk patients. Crit Care. 2013 Feb 28;17(1):R35. doi: 10.1186/cc12544. PMID 23448570
- [Background] Fuster-Lluch O, Geronimo-Pardo M, Peyro-Garcia R, Lizan-Garcia M. Glomerular hyperfiltration and albuminuria in critically ill patients. Anaesth Intensive Care. 2008 Sep;36(5):674-80. doi: 10.1177/0310057X0803600507. PMID 18853585
- [Background] Udy AA, Roberts JA, Boots RJ, Paterson DL, Lipman J. Augmented renal clearance: implications for antibacterial dosing in the critically ill. Clin Pharmacokinet. 2010;49(1):1-16. doi: 10.2165/11318140-000000000-00000. PMID 20000886
- [Background] Claus BO, Hoste EA, Colpaert K, Robays H, Decruyenaere J, De Waele JJ. Augmented renal clearance is a common finding with worse clinical outcome in critically ill patients receiving antimicrobial therapy. J Crit Care. 2013 Oct;28(5):695-700. doi: 10.1016/j.jcrc.2013.03.003. Epub 2013 May 14. PMID 23683557
- [Background] Minkute R, Briedis V, Steponaviciute R, Vitkauskiene A, Maciulaitis R. Augmented renal clearance--an evolving risk factor to consider during the treatment with vancomycin. J Clin Pharm Ther. 2013 Dec;38(6):462-7. doi: 10.1111/jcpt.12088. Epub 2013 Aug 8. PMID 23924288
- [Background] Cook AM, Arora S, Davis J, Pittman T. Augmented renal clearance of vancomycin and levetiracetam in a traumatic brain injury patient. Neurocrit Care. 2013 Oct;19(2):210-4. doi: 10.1007/s12028-013-9837-y. PMID 23907742
- [Background] Udy AA, Varghese JM, Altukroni M, Briscoe S, McWhinney BC, Ungerer JP, Lipman J, Roberts JA. Subtherapeutic initial beta-lactam concentrations in select critically ill patients: association between augmented renal clearance and low trough drug concentrations. Chest. 2012 Jul;142(1):30-39. doi: 10.1378/chest.11-1671. PMID 22194591